CLINICAL TRIAL: NCT06603415
Title: Pattern of Hashimoto's Thyroiditis in Upper Egypt
Brief Title: Hashimoto's Thyroiditis in Upper Egypt
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Hossam Mohamed Araby, Resident, Department of General Surgery, Faculty of Medicine, Sohag University, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-24-07-06MS
Record Dates: First submitted 2024-08-29; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Hashimoto's Thyroiditis
MeSH Terms: conditions — Hashimoto Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PATTERN OF HASHIMOTO'S THYROIDITIS IN UPPER EGYPT (Other): the pathological pattern, characteristics, treatment, complications and prognosis of Hashimoto's thyroiditis in upper egypt .
  Interventions: Procedure: Total thyroidectomy

INTERVENTIONS:
Procedure: Total thyroidectomy — Total thyroidectomy (with preservation of bilateral recurrent laryngeal nerves and all parathroid glands) for histopathology

SUMMARY:
The aim of this study is to evaluate the pathological pattern, characteristic features, treatment, complications and prognosis of Hashimoto's thyroiditis in upper Egypt.

ELIGIBILITY:
Inclusion Criteria:

* All patients with Hashimoto's thyroiditis, males or females, any age, at upper egypt .

Exclusion Criteria:

* Patients with associated other thyroid pathology other than Hashimoto's thyroiditis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Early post operative follow up of Hashimoto's thyroiditis | 3 days after the operation
  Removal of suction drains

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Sohag University Hospital, Sohag
  - Sohag university hospital, Sohag

REFERENCES:
- [Background] Feldt-Rasmussen U. Hashimoto's thyroiditis as a risk factor for thyroid cancer. Curr Opin Endocrinol Diabetes Obes. 2020 Oct;27(5):364-371. doi: 10.1097/MED.0000000000000570. PMID 32773575
- [Background] Cipolla C, Sandonato L, Graceffa G, Fricano S, Torcivia A, Vieni S, Latteri S, Latteri MA. Hashimoto thyroiditis coexistent with papillary thyroid carcinoma. Am Surg. 2005 Oct;71(10):874-8. PMID 16468540
- [Background] Kashima K, Yokoyama S, Noguchi S, Murakami N, Yamashita H, Watanabe S, Uchino S, Toda M, Sasaki A, Daa T, Nakayama I. Chronic thyroiditis as a favorable prognostic factor in papillary thyroid carcinoma. Thyroid. 1998 Mar;8(3):197-202. doi: 10.1089/thy.1998.8.197. PMID 9545105